CLINICAL TRIAL: NCT04955665
Title: The Clinical Efficacy of Reattachment of the Superior Peroneal Retinaculum Versus the Bone Block Procedure for Recurrent Peroneal Tendon Dislocation
Brief Title: Reattachment of the SPR Versus the Bone Block Procedure for Recurrent Peroneal Tendon Dislocation
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2018225
Record Dates: First submitted 2021-06-25; First posted 2021-07-09 (Actual); Last update posted 2021-07-09 (Actual); Status verified 2021-06

CONDITIONS: Recurrent Peroneal Tendon Dislocation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Bone block procedure: patients with recurrent peroneal tendon dislocation underwent the bone block procedure
  Interventions: Procedure: bone block procedure
- Reattachment of the superior peroneal retinaculum: patients with recurrent peroneal tendon dislocation underwent reattachment of the superior peroneal retinaculum
  Interventions: Procedure: Reattachment of the superior peroneal retinaculum

INTERVENTIONS:
Procedure: bone block procedure — a 20 × 15 × 3 mm3 bone block was cut from the lateral malleolus, rotated backwards 45°, and sutured back to the periosteum of the lateral malleolus using non-absorbable sutures.
  Groups: Bone block procedure
Procedure: Reattachment of the superior peroneal retinaculum — two suture anchors (Mini Quickanchor,DePuy Mitek) were inserted into the postero-lateral ridge of the lateral malleolus without damaging the cartilaginous ridge, after which the SPR was reattached to the lateral malleolus with the anchored suture. The inner layer of the false pouch was incised, and the outer layer (periosteum) was sutured with the SPR in a pants-over-vest style.
  Groups: Reattachment of the superior peroneal retinaculum

SUMMARY:
Clinical outcomes between reattachment of the superior peroneal retinaculum (SPR) and the bone block procedure were compared in this study to elucidate which procedure was safer and more effective.

DETAILED DESCRIPTION:
From 2012 to 2016, 25 patients with recurrent peroneal tendon dislocation underwent the bone block procedure(group A), and another 22 patients underwent reattachment of the SPR (group B). American Orthopaedic Foot and Ankle society (AOFAS) ankle-hindfoot score, Ankle Activity Score (AAS), time to return to sports activity, rate of return to sports level, range of motion (ROM) of the ankle, rate of recurrence, and overall patient satisfaction were collected to evaluate outcomes between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* a traumatic recurrent peroneal tendon dislocation requiring surgery
* a lack of response to at least 3 months of conservative treatment

Exclusion Criteria:

* the presence of an acute peroneal tendon dislocation
* a concomitant anterior talofibular ligament rupture

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A consecutive series of patients with recurrent peroneal tendon dislocation who underwent operative treatment between 2012 and 2016 were retrieved. Twenty-five patients underwent bone block procedure (group A), and 22 patients underwent reattachment of the SPR (group B)."
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2012-07-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
AOFAS | 2 years after operation
  The American Orthopaedic Foot and Ankle Society (AOFAS) Ankle-Hindfoot Score combines subjective scores of pain and function provided by the patient with objective scores based on the surgeon's physical examination of the patient (to assess sagittal motion, hindfoot motion, ankle-hindfoot stability and alignment of the ankle-hindfoot). The scale includes nine items that can be divided into three subscales (pain, function and alignment). The minimum and maximum values of AOFAS are 100 and 0, respectively. And higher scores mean a better outcome.

SECONDARY OUTCOMES:
VAS | 2 years after operation
  The Visual Analogue Scale (VAS) is designed to present to the respondent a rating scale with minimum constraints. Respondents mark the location on the 10-centimeter line corresponding to the amount of pain they experienced. This gives them the greatest freedom to choose their pain's exact intensity. It also gives the maximum opportunity for each respondent to express a personal response style. The minimum and maximum values of VAS are 10 and 0, respectively. And higher scores mean a worse outcome.
time to return to sports activity | up to 2 years
  time to return to sports activity after surgery at each group

CONTACTS AND LOCATIONS:
Overall Officials: Qinwei Guo, MD, Study Chair — Peking University Third Hospital

IPD SHARING:
Plan to Share IPD: No